CLINICAL TRIAL: NCT01368029
Title: Double Blind Randomized Controlled Trial to Evaluate the Safety of Lactobacillus Rhamnosus GG ATCC 53103 (LGG) Vs. Placebo in Elderly Subjects Receiving Trivalent Inactivated Influenza Vaccine
Brief Title: Safety of Lactobacillus Rhamnosus GG Vs. Placebo in Elderly Subjects Receiving Trivalent Inactivated Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia L. Hibberd, Chief; Division of Global Health; MGHfC, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2010 P 001694
Record Dates: First submitted 2011-06-02; First posted 2011-06-07 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Healthy; Elderly
Keywords: LGG; Immune response; Influenza vaccine; Elderly; Healthy; Microbiome
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LGG (Experimental): Lactobacillus rhamnosus GG (LGG) containing 1x10^10 LGG per capsule will be given to volunteers with verbal and written instructions at the baseline visit. Capsules are to be taken orally twice a day on an outpatient basis.
  Interventions: Biological: Lactobacillus rhamnosus GG ATCC 53103 (LGG)
- Placebo (Placebo Comparator): Placebo capsules composed of microcrystalline cellulose are to be taken orally twice a day on an outpatient basis.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus rhamnosus GG ATCC 53103 (LGG) — Study drug capsules (1x10^10 LGG/capsule) are to be taken orally twice a day every day on an outpatient basis for 28 days
  Other Names: Culturelle; LGG
  Arms: LGG
Biological: Placebo — Placebo capsules composed of microcrystalline cellulose are to be taken orally twice a day on an outpatient basis for 28 days.
  Arms: Placebo

SUMMARY:
This is a phase I, randomized controlled trial to evaluate the safety of Lactobacillus rhamnosus GG (LGG) versus placebo in elderly subjects receiving the trivalent inactivated influenza vaccine. Lactobacilli are part of the normal flora of the intestine. LGG is one of several strains of Lactobacilli that is used as a probiotic or microorganism administered to confer "health benefits". Our research is focused on studying the possible therapeutic effects of LGG. The study hypotheses are:

1. LGG or placebo administered twice daily will be safe and well tolerated in elderly subjects who have just received the trivalent inactivated influenza vaccine
2. The immune response to the influenza vaccine at day 21, 28, 56, and at the end of the influenza season will be higher in the LGG group than the placebo group
3. The occurrence rate of influenza like illness during the influenza season will be lower in the LGG group than in the placebo group
4. The diversity of the microbiota in nasopharyngeal and stool specimens at day 21, 28, 56 and at the end of the influenza season will be greater in the LGG group than the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-80 years
2. Willing to complete the informed consent process
3. Able and willing to participate for the planned duration of the study, including availability for follow-up telephone contact
4. Is community dwelling for the past two years
5. Has received routine physical in the past two years
6. Has no new chronic conditions in the past two years
7. Identifies a primary care clinician
8. Has received recommended preventive services (Task Force for Clinical Preventive Services) for vaccination and cancer prevention/detection, e.g.:

   1. Pneumococcal vaccination
   2. Mammography
   3. Screening colonoscopy for cancer
9. Willing to comply with protocol and report on compliance and side effects during the study period
10. Informed consent obtained and signed prior to screening

Exclusion Criteria:

1. Self-reported vaccination with influenza vaccine for the current season
2. Vaccination with any vaccine within the one month period prior to study enrollment or intent to receive any other vaccine during the study period
3. History of hypersensitivity to any influenza vaccine components including thimerosal or egg
4. History of Guillain-Barre syndrome
5. History of avoidance of egg and/or egg based products for any reason
6. Acute febrile illness within the week prior to immunization - immunization deferred until illness resolved
7. Consumption of supplements or food products containing LGG or probiotics for 28 days prior to the start of the study or consumption of yogurt that has the "live and active cultures" seal
8. Known or suspected allergies to probiotics, Lactobacillus, microcrystalline cellulose, gelatin, or antibiotics that may be used to treat LGG bacteremia or infection
9. Received oral or parenteral antibiotics within 4 weeks of enrollment or prescribed antibiotics on the day of enrollment
10. Drug or alcohol abuse within the previous 12 months
11. Hospitalization, major surgery or endoscopy within the last 3 months
12. Scheduled hospital admission within 3 months of enrollment
13. Resident of a nursing home or rehabilitation center
14. Presence of any of the following:

    1. Grade 2 or higher abnormal vital signs or abnormalities on physical exam
    2. Indwelling catheter or implanted hardware/prosthetic device or feeding tube
    3. Current or within the last 2 years, any episode of bowel leak, acute abdomen, diverticulitis, bloody bowel movements or peptic ulcer disease, including any surgical procedure or current prescription medications for any of these conditions
    4. Current or within the last 4 weeks, active bowel disease such as an episode of infectious or non-infectious diarrhea, constipation or vomiting lasting more than 12 hours or current prescription medications for any of these conditions
    5. Any history of gastric or intestinal dysmotility, slowed transit time, variable small intestinal permeability, pancreatitis, history of disease or current prescription medication for any of these conditions
    6. Any history of Hepatitis B or Hepatitis C infections, cirrhosis, or chronic liver disease
    7. Underlying structural heart disease such as abnormal native heart valve replacement, Stage IV congestive heart failure
    8. History of peripheral vascular disease or stroke
    9. Immunosuppression including HIV positive, solid organ or stem cell transplant recipient, receiving any oral or parenteral immunosuppressive therapy, neutrophil count <500/mm^3, or an anticipated drop in the neutrophil count to <500/mm^3 or active or planned chemotherapy or radiotherapy
    10. History of collagen vascular or autoimmune disease
    11. End stage renal disease
    12. History of chronic obstructive pulmonary disease or asthma
    13. Diabetes or thyroid disease
    14. Active tuberculosis (TB), defined as undergoing a work up for suspected active TB infection or currently on treatment for active TB
15. Positive drug or alcohol testing at screening or positive breathalyzer at baseline or an unwillingness to undergo drug and alcohol testing
16. Abnormal laboratory tests defined as any of the following:

    1. White blood cell (WBC) <3.3 or > 12.0 K/microliter
    2. Platelets < 125 K/microliter
    3. Hemoglobin Males: < 12.0 g/dL; Females < 11.0 g/dL
    4. Creatinine > 1.8 mg/dL
    5. Blood Urea Nitrogen (BUN)> 27 mg/dL
    6. Aspartate aminotransferase (AST) > 1.25 ULN
    7. Alanine aminotransferase > 1.25 ULN
    8. Alkaline phosphatase > 2.0 ULN
    9. Bilirubin (total) > 1.5 ULN
    10. Glucose (nonfasting) > 126 mg/dL
    11. Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody
17. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the subject participating in the study or would make it unlikely the subject could complete the study

    -

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events that are possibly or probably related to administration of LGG | Subjects will be followed from the study start through the end of the influenza season (as defined by CDC) with an anticipated average for most subjects of 7 months.
  Adverse events will be detected during study visits with standardized questionnaires, medical history, vital signs, physical examinations, laboratory tests and review of subject diaries as well as between study visits on telephone calls based on responses to adverse event questionnaires. Additionally, subjects are encouraged to call the PI or study staff at any time if they are experiencing an adverse event.

SECONDARY OUTCOMES:
Anti-influenza systemic immune response | Subjects will be followed from the study start through the end of the influenza season (as defined by CDC) with an anticipated average for most subjects of 7 months.
  HAI, MN titers and IgA titers will be measured at days 21, 28, 56 and the end of the influenza season
Anti-influenza mucosal immune response | Subjects will be followed from the study start through the end of the influenza season (as defined by CDC) with an anticipated average for most subjects of 7 months.
  IgA titers will be measured at days 21, 28, 56 and at the end of the influenza season
Occurrence of influenza like illness | Subjects will be followed from the study start through the end of the influenza season (as defined by CDC) with an anticipated average for most subjects of 7 months.
  Influenza like illness is defined as a reported oral temperature of 100 degrees Fahrenheit with at least 2 symptoms of acute respiratory illness
Changes in the richness and bacterial diversity of the nasopharyngeal and gut microbiota and presence of LGG in stool specimens by routine culture | Subjects will be followed from the study start through the end of the influenza season (as defined by CDC) with an anticipated average for most subjects of 7 months.
  Stool and nasopharyngeal specimens will be analyzed to learn what bacteria are present during different phases of the study and how the types and quantities of bacteria may change over time

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L. Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States